CLINICAL TRIAL: NCT05844722
Title: Effectiveness of Mindfulness-based Cognitive Therapy Undergoing Post-stroke Rehabilitation: a Randomized Controlled Trial
Brief Title: Effectiveness of Mindfulness-based Cognitive Therapy Undergoing Post Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Medical Rehabilitation, Hungary (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60371-2/2018/EKU
Record Dates: First submitted 2023-04-03; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Rehabilitation; Mindfulness
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCT group (Experimental): The intervention group were involved in MBCT intervention in addition to usual care. MBCT intervention was designed to consist of eight 1.5-hour group sessions over 6 consecutive weeks.
  Interventions: Behavioral: Mindfulness-based intervention therapy
- Control group (Active Comparator): Received usual care (standard multidisciplinary stroke care) over 6 weeks.
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: Mindfulness-based intervention therapy — Mindfulness-based cognitive therapy consists of meditation techniques to stay in the present moment with acceptance (breathing exercises, body scan, gentle yoga, awareness of thoughts and feelings) and some aspects of cognitive therapy, and psycho-education.
  Arms: MBCT group
Other: usual care — Usual care means received standard multidisciplinary stroke care
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of mindfulness-based cognitive therapy compared to usual care for stroke survivors undergoing inpatient rehabilitation.

DETAILED DESCRIPTION:
It was hypothesized that group-based MBCT would lead to improving mood, mindfulness, social support, physical, and neurocognitive function; and that these improvements would be maintained over the 3-month follow-up period. Participants in the control group received only usual care, the intervention group were involved in MBCT intervention in addition to usual care. MBCT intervention was designed to consist of eight 1.5-hour group sessions over 6 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* stroke patients with functional impairments
* confirmation of stroke by CT or MRI scan
* age between 18-90 years
* had adequate communication skills, cognitive and physical capacity to participate in study activities
* competence to provide informed consent

Exclusion Criteria:

* severe cognitive impairment according to the Word List Learning Instrument (total score <7)
* severe depression according to the Beck Depression Inventory (BDI) (total score>25)
* history of severe mental illness (psychotic disorder, schizophrenia, severe depression, bipolar disorder, PTSD, suicidal tendencies)
* the current change in the antidepressant therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Beck Depression Inventory (BDI) at 6 weeks | Baseline and 6 weeks
  Beck Depression Inventory (BDI) was used to assess severity of the depression with 21 items scored from 0 to 3 (hiv, Beck, 1961). Scores range from 0 to 63 with 0-9 representing normal value, 10-18 mild, 19-25 moderate, and ≥ 26 severe depression.
Change from 6 weeks on Beck Depression Inventory (BDI) at 3 months | 6 weeks and 3 months
  Beck Depression Inventory (BDI) was used to assess severity of the depression with 21 items scored from 0 to 3 (hiv, Beck, 1961). Scores range from 0 to 63 with 0-9 representing normal value, 10-18 mild, 19-25 moderate, and ≥ 26 severe depression.
Change from baseline on The Spielberger State-Trait Anxiety Inventory (STAI-X) at 6 weeks | Baseline and 6 weeks
  The Spielberger State-Trait Anxiety Inventory (STAI-X) was used to assess anxiety both as a state and trait. State anxiety was measured by STAI form X-1, requiring participants to answer questions about how they feel right now. Trait anxiety was measured by the STAI form X-2, requiring participants to answer questions about how they feel generally. Both scales (X-1, X-2) consist of 20 items scored from 1 to 4. Scores range from 20 to 80 with higher scores representing higher state or trait anxiety.
Change from 6 weeks on The Spielberger State-Trait Anxiety Inventory (STAI-X) at 3 months | 6 weeks and 3 months
  The Spielberger State-Trait Anxiety Inventory (STAI-X) was used to assess anxiety both as a state and trait. State anxiety was measured by STAI form X-1, requiring participants to answer questions about how they feel right now. Trait anxiety was measured by the STAI form X-2, requiring participants to answer questions about how they feel generally. Both scales (X-1, X-2) consist of 20 items scored from 1 to 4. Scores range from 20 to 80 with higher scores representing higher state or trait anxiety.

SECONDARY OUTCOMES:
Change from baseline on The Five Facet Mindfulness Questionnaire (FFMQ) at 6 weeks | Baseline and 6 weeks
  Five Facet Mindfulness Questionnaire (FFMQ) was used to assess mindfulness with 39 items scored from 1 to 5 with five subscales, including observing (8 items), describing (8), acting with awareness (8), nonjudging of inner experience (8), and nonreactivity to inner experience (7). Total scores range from 39 to 195 with higher scores representing higher mindfulness.
Change from 6 weeks on The Five Facet Mindfulness Questionnaire (FFMQ) at 3 months | 6 weeks and 3 months
  Five Facet Mindfulness Questionnaire (FFMQ) was used to assess mindfulness with 39 items scored from 1 to 5 with five subscales, including observing (8 items), describing (8), acting with awareness (8), nonjudging of inner experience (8), and nonreactivity to inner experience (7). Total scores range from 39 to 195 with higher scores representing higher mindfulness.
Change from baseline on The Multidimensional Scale of Perceived Social Support Scale(MSPSS) at 6 weeks | Baseline and 6 weeks
  Multidimensional Scale of Perceived Social Support (MSPSS) was used to assess perceived social support receives from 3 different sources: family, friends, and significant other. The original version of the MSPSS is a 12-item scale scored from 0 to 6. The validated Hungarian version consists of 10 items scored from 1 to 5. Scores range from 10 to 50 with higher scores representing higher perceived social support.
Change from 6 weeks on The Multidimensional Scale of Perceived Social Support Scale (MSPSS) at 3 months | 6 weeks and 3 months
  Multidimensional Scale of Perceived Social Support (MSPSS) was used to assess perceived social support receives from 3 different sources: family, friends, and significant other. The original version of the MSPSS is a 12-item scale scored from 0 to 6. The validated Hungarian version consists of 10 items scored from 1 to 5. Scores range from 10 to 50 with higher scores representing higher perceived social support.
Change from baseline on Touluose-Piéron test(TP) at 6 weeks | Baseline and 6 weeks
  Touluose-Piéron (TP) was used to assess sustained attention. This paper-pencil test consists of small boxes that have lines oriented in different directions, distributed in columns and rows. The task of the test is to examine the boxes and to mark those matching 4 model boxes, as quickly as possible within a limited time. Noted scores: the number of correct answers (CA), errored boxes (E), and omitted boxes (O). The Global Index of Attention and Perception (GIAP) is calculated by: CA- (E + O). Higher scores represent higher sustained attention.
Change from 6 weeks on Touluose-Piéron test(TP) at 3 months | 6 weeks and 3 months
  Touluose-Piéron (TP) was used to assess sustained attention. This paper-pencil test consists of small boxes that have lines oriented in different directions, distributed in columns and rows. The task of the test is to examine the boxes and to mark those matching 4 model boxes, as quickly as possible within a limited time. Noted scores: the number of correct answers (CA), errored boxes (E), and omitted boxes (O). The Global Index of Attention and Perception (GIAP) is calculated by: CA- (E + O). Higher scores represent higher sustained attention.
Change from baseline on Fugl-Meyer Assessment (FMA) at 6 weeks | Baseline and 6 weeks
  Fugl-Meyer Assessment (FMA) is a clinician-measured instrument used to assess sensorimotor impairment in patients with post-stroke. It assess motor functioning, sensation, balance, joint range of motion and joint pain. The current study applied only the domain of the motor function (in the upper and lower extremities), and balance. The 57 items scored on a 3-point ordinal scale from 0 to 2, with a higher score representing less impairment. The motor score (M) ranges from 0 to 100; upper extremity (UE) 33 items with scores ranging from 0 to 66, lower extremity (LE) 17 items with scores ranging from 0 to 34. Balance 7 items scores from 0 to 14.
Change from 6 weeks on Fugl-Meyer Assessment (FMA) at 3 months | 6 weeks and 3 months
  Fugl-Meyer Assessment (FMA) is a clinician-measured instrument used to assess sensorimotor impairment in patients with post-stroke. It assess motor functioning, sensation, balance, joint range of motion and joint pain. The current study applied only the domain of the motor function (in the upper and lower extremities), and balance. The 57 items scored on a 3-point ordinal scale from 0 to 2, with a higher score representing less impairment. The motor score (M) ranges from 0 to 100; upper extremity (UE) 33 items with scores ranging from 0 to 66, lower extremity (LE) 17 items with scores ranging from 0 to 34. Balance 7 items scores from 0 to 14.
Change from baseline on Functional Independence Measure (FIM) at 6 weeks | Baseline and 6 weeks
  Functional Independence Measure (FIM) was used to assess the level of independence in basic activities of daily living. FIM is a clinician-measured instrument consisting of 13 motor and 5 cognitive items scored from 1 to 7. The higher the score, the more independent the patient. Scores from 1 to 5 indicate a need for assistance. The total score ranges from 18 and 126; the motor subscale score ranges from 13 to 91, and the cognitive subscale score ranges from 5 to 35.
Change from 6 weeks on Functional Independence Measure (FIM) at 3 months | 6 weeks and 3 months
  Functional Independence Measure (FIM) was used to assess the level of independence in basic activities of daily living. FIM is a clinician-measured instrument consisting of 13 motor and 5 cognitive items scored from 1 to 7. The higher the score, the more independent the patient. Scores from 1 to 5 indicate a need for assistance. The total score ranges from 18 and 126; the motor subscale score ranges from 13 to 91, and the cognitive subscale score ranges from 5 to 35.

CONTACTS AND LOCATIONS:
Overall Officials: Gábor Fazekas, MD habil PhD, Principal Investigator — National Institute for Medical Rehabilitation, Hungary
Locations (1):
- National Institute for Medical Rehabilitation, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No